CLINICAL TRIAL: NCT04054401
Title: SynerFuse Spinal Fusion and Neuromodulation Proof of Concept Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SynerFuse, Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G190045
Record Dates: First submitted 2019-07-30; First posted 2019-08-13 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Spinal Fusion; Radiculopathy Lumbar; Chronic Pain
Keywords: Dorsal Root Ganglion; Neurostimulation; Failed Back Surgery Syndrome
MeSH Terms: conditions — Chronic Pain; Failed Back Surgery Syndrome | interventions — Spinal Fusion

STUDY DESIGN:
Intervention Model Description: Single group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- DRG Neurostimulation with Spinal Fusion (Experimental)
  Interventions: Device: DRG Neurostimulation with Spinal Fusion

INTERVENTIONS:
Device: DRG Neurostimulation with Spinal Fusion — Surgeons will implant a neurostimulator during the same open back procedure as fusion devices (spinal fusion hardware and interbody cage) and begin neurostimulation in a short time following surgery (24 hours).

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of DRG stimulation when placing a neurostimulator during the same procedure as implantation of spinal fixation with or without interbody cage systems in patients with chronic back and/or leg pain requiring single level spinal fusion.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for a single level or two level adjacent spinal fusion having back pain and radiculopathy
* Have been diagnosed with chronic, intractable pain of the lower back and/or leg refractory to conservative therapy for at least 3 of months
* At least 6 months since last surgical procedure on the spine
* Be 21 years of age or older at the time of enrollment
* Be willing and capable of giving informed consent
* Be willing and able to comply with study-related requirements

Exclusion Criteria:

* Any prior spinal fusion at index or adjacent level
* Pregnant
* Have a life expectancy of less than 1 year
* Be concomitantly participating in another clinical study
* Be involved in an injury claim under current litigation
* Baseline narcotic use of ≥ 100 MME per day
* Significant untreated addiction to dependency producing medications
* Current active implantable medical device
* Cancer
* Have osteoporosis
* Active infection
* Allergies to system components
* AGE > 80
* Expected need to undergo MRI imaging in the future
* Other significant comorbidities

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Characterization of device-related adverse events | Surgery through 12 months post-op
Primary Effectiveness Endpoint: Change in back and leg pain Visual Analog Score (VAS) scores | Baseline to 3 months post-op
  VAS scores range from 0 (no pain) to 100 (pain is as bad as it could possibly be). Decreases in scores indicate reductions in pain.

SECONDARY OUTCOMES:
Change in neurological status | Baseline to 3, 6, and 12 months post-op
  Change in neurological status measured by the neurological component of the standard physical exam.
Change in disability measured by the Oswestry Disability Index (ODI). | Baseline to 3, 6, and 12 months post-op
  Each question is scored from 0-5. The scores from each question are summed, then divided by the maximum number possible, then multiplied by 100 to represent a percentage. The percentages are broken down into 5 category ranges: 0% to 20%: minimal disability, 21%-40%: moderate disability; 41%-60%: severe disability; 61%-80%: crippled; 80%-100%: bed-bound or exagerating.
Change in quality of life as measured by PROMIS Scale v1.2 - Global Health. | Baseline to 3, 6, and 12 months post-op
  The is a 10-item patient-reported questionnaire in which the response options are presented as a 5-point rating scale. The results of the scores are are used to calculate two summary scores: a Global Physical Health score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score." The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
Change in quality of life as measured by EQ-5D-5L. | Baseline to 3, 6, and 12 months post-op
  The EQ-5D-5L survey consists of 5 dimensions with the score for each ranging from 1 (no problems) to 5 (unable to do). For individual dimensions, negative changes (e.g. from 5 to 3) indicate improvement. The scores on these five dimensions will be presented as a health profile and converted to a single summary index number (utility). Positive changes in the total score indicate improvement.
Change in use of analgesics over time | Baseline through 12 months post-op
  Change in use of medications at all follow up visits.

OTHER OUTCOMES:
Amount of device migration | Surgery to 3, 6, and 12 months post-op
  Amount of device migration as measured by anteroposterior (AP) and lateral x-rays.
Costs and cost-effectiveness of the intervention | Baseline through 12 months post-op
  The cost effectiveness analysis will report total healthcare-related expenditures reported by patients from baseline to 12 months post-op and 12 month quality-adjusted life-years (QALYs). Incremental cost per QALY will be estimated and compared to previously published studies.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - South Bend Orthopaedics, Mishawaka, Indiana
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No
There are no plans to make the IPD available to other researchers.